CLINICAL TRIAL: NCT00744653
Title: Electrochemotherapy for Chest Wall Recurrence af Breast Cancer: Present Challenges and Future Prospects.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Primary endpoint measure not suitable for evaluation
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-B-2008-074
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Results first posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-06

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Recurrence
MeSH Terms: conditions — Breast Neoplasms; Recurrence | interventions — Electrochemotherapy; Bleomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Patients with local-regional recurrence of breast cancer, lesion over 3 cm.
  Interventions: Procedure: Electrochemotherapy

INTERVENTIONS:
Procedure: Electrochemotherapy — Electric pulses , duration 100 microseconds, about 400 V given at 5000 Hz. Drug used is Bleomycin.
  Other Names: Device: Cliniporator; Drug: Bleomycin

SUMMARY:
By applying short electric pulses to cells, the cell membranes can become permeabilised (electroporation). This can be used augment the effect of chemotherapy, by providing direct access to the cell cytosol. For the drug bleomycin, the enhancement of effect is several hundred fold, enabling once-only treatment. We wish to offer electrochemotherapy to breast cancer patients suffering from chest wall recurrences that are ulcerated or painful and where other treatments have failed.

DETAILED DESCRIPTION:
Electrochemotherapy for chest wall recurrence of breast cancer. MD, Ph.D. student, Louise Wichmann Matthiessen, has been employed in 2008 to perform this study. She plans to complete her training as specialist in clinical oncology subsequently, and will thus be able to follow up the work after completion of her Ph.D. The study aims at giving palliation to patients who are suffering from painful, ulcerated metastases to the chest wall in a situation where other treatments have failed.

Inclusion criteria: Chest wall recurrence of breast cancer; all other modalities have failed or patients does not wish to receive them (e.g. chemotherapy); symptomatic relief is needed; WHO performance status 0-2; normal coagulation parameters, normal kidney and renal function; written, informed consent. Lesions totalling over 3 cm in diameter. Patient recruitment: 28 patients are to be recruited.

Treatment: Patients will be treated in general anesthesia (inhaling max. 30 % oxygen), and a standard dose of bleomycin (15.000 IU/ m2) will be given intravenously. Electric pulses will be administered using a square wave electroporator (IGEA, Carpi, Italy). Needle and plate electrodes are used in order to treat the affected area efficiently. Eight pulses at a frequency of 5 kHz will be used for each application of the electrodes. In this way, a large area can be treated within a short time. Post treatment, the area will be covered by dry dressings, as are standardly used.

The patients will be seen at 2, 4, and 8 weeks post treatment, and re-treatment can be administered up to three times in case there are areas which have not been insufficiently treated in the first round. Lung function will be followed by measurement of DLCO (carbon monoxide diffusion capacity).

The patients will furthermore be followed up to 1 year after treatment in monthly intervals, and after 1 year on a yearly basis for up to 5 years.

Evaluation: Evaluation is performed by a) measurement of lesion extension and digital photography, b) development of a mapping system: Chest wall recurrences are frequently a confluent mass of tumor with varying depth. Precise mapping of treatment areas and effect is warranted. To this end, a system combining a fixed point (e.g. small ink tattoo, as used in radiotherapy planning) with novel imaging techniques using the 3D computer tomography (CT) planning system employed for radiotherapy, is envisaged. Furthermore, PET-Dual Time Point scanning combined with CT scanning is being investigated as treatment evaluation.

Safety: Safety will be reported both in terms of evaluation of adverse events and in terms of patient satisfaction determined by questionnaire, including the 'Derriford Appearance Questionaire'(18).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Histological proven cancer of the breast.
* Progressive and/or metastatic disease.
* No further standard treatment for the patient available or the patient does not wish to receive the offered standard treatment.
* If Endocrine therapy: Progression in cutaneous lesions.
* If treatment with trastuzumab (Herceptin)can continue this treatment if there is no regression in cutaneous lesions.
* At least 2 weeks since last chemotherapy, patients treated with Navelbine (Vinorelbine), Capecitabin (Xeloda) or weekly Paclitaxel (Taxol)can continue this treatment if there is no regression in cutaneous metastases.
* Malignant cutaneous or subcutaneous lesion to be treated ≥ 3 cm.
* WHO performance ≤ 2.
* Life expectancy of at least 3 months.
* Platelets ≥ 50 mia/l, pp ≥ 40, APTT in normal area. Medical correction is allowed.
* Sexual active men and women must use safe anticonceptive during and up to 6 month after last treatment.
* Written informed consent must be obtained according to the local Ethics committee requirements.

Exclusion Criteria:

* Acute lung infection
* Previous bleomycin treatment exceeding 200.000 Units/m2.
* Known hypersensitivity to any of the components of the treatment.
* Known hypersensitivity to any of the components used in the planned anesthesia.
* Pregnant or lactating women. In fertile women this is ensured by measuring HCG in blood.
* Treatment with granulocyte colony stimulating factor (G-CSF) or other cytokines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-10; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Gehl, M.D., Principal Investigator — Department of Oncology, Copenhagen University Hospital at Herlev
Locations (1):
- Herlev Hospital, Herlev Ringvej 75, Herlev, Denmark

REFERENCES:
- [Result] Matthiessen LW, Johannesen HH, Hendel HW, Moss T, Kamby C, Gehl J. Electrochemotherapy for large cutaneous recurrence of breast cancer: a phase II clinical trial. Acta Oncol. 2012 Jul;51(6):713-21. doi: 10.3109/0284186X.2012.685524. Epub 2012 Jun 26. PMID 22731832

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment period: October 2008 to November 2010. Total of 17 patients included and treated with electrochemotherapy.
Groups:
- Electrochemotherapy: Patients with local-regional recurrence of breast cancer, lesion over 3 cm. Treatment with electric pulses combined with bleomycin. Pulse duration 100 microseconds, about 400 V given at 5000 Hz.
Period: Overall Study
Arm/Group | Electrochemotherapy
Started | 17
Completed | 1
Not Completed | 16
Not completed — antineoplastic treatment | 11
Not completed — Death | 1
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | Electrochemotherapy
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 0
Region of Enrollment [Number; unit: participants]
  Denmark | 17

OUTCOME MEASURES:

1. Primary Outcome: Clinical Measure of Lesion Size.
Description: Response was evaluated clinical using Response Evaluation Criteria in Solid Tumors (RECIST) guidelines and documented with digital photography. Number of patients with objective response evaluated with clinical measure of lesion size
Time Frame: up to one year
Population: Based on Simons optimal design for phase II trials, 25 evaluable patients were to be included and treated.
Measure: Number; unit: Participants
Arm/Group | Electrochemotherapy
Number analyzed (Participants) | 12
Participants | 2

2. Secondary Outcome: Participants With Objective Response Evaluated With PET/CT
Description: Participants with objective response evaluated with PET/CT. Objective Response evaluated with CT and PET/CT.
Time Frame: 3, weeks, 8 weeks, and up to 6 months after treatment
Population: per protocol
Measure: Number; unit: participants
Groups:
- Electrochemotherapy: All patients treated with electrochemotherapy
Arm/Group | Electrochemotherapy
Number analyzed (Participants) | 12
participants | 4

3. Secondary Outcome: Safety and Toxicity
Time Frame: up to 1 year
Population: per protocol
Measure: Number; unit: adverse events
Units Other Than Participants: number of adverse events
Arm/Group | Electrochemotherapy
Number analyzed (Participants) | 16
Number analyzed (number of adverse events) | 0
adverse events | 0

ADVERSE EVENTS:
Arm/Group | Electrochemotherapy
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

LIMITATIONS AND CAVEATS:
Early termination due to too few objective respondes using the primary endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes